CLINICAL TRIAL: NCT07286604
Title: Repurposing Ivermectin (IVM) for Treatment of Post Kala-azar Dermal Leishmaniasis (PKDL): Safety and Response to Multiple Doses of Ivermectin
Brief Title: Ivermectin Repurposed for the Treatment of PKDL
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR-21134
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Post Kala Azar Dermal Leishmaniasis
MeSH Terms: interventions — Ivermectin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tablet Ivermectin (Experimental)
  Interventions: Drug: Ivermectin 6 MG Oral Tablet (2 tablets)

INTERVENTIONS:
Drug: Ivermectin 6 MG Oral Tablet (2 tablets) — A cumulative dose of 60 mg Oral Ivermectin monotherapy (12 mg/day) on five consecutive days (day 1 - day 5) for three consecutive months (180 mg in total)

SUMMARY:
Background (brief):

1. Burden: Post-Kala-Azar Dermal Leishmaniasis (PKDL) commonly follows visceral leishmaniasis (VL) caused by Leishmania donovani. It is characterized by skin lesions in which parasites can be identified, in a patient who is otherwise fully recovered from VL or exposed to L. donovani (LD) infection. It occurs in the Indian subcontinent (mainly India and Bangladesh) as well as in Africa (mainly Sudan). It is now established that PKDL patients play an important role in transmission of LD parasite where chronic PKDL patients have been implicated in major VL outbreaks in the past. In a series of cross-sectional surveys between 2002-2010, the cumulative incidence of PKDL was estimated at 17% by 5 years in Bangladesh. Most patients had been treated with SSG (95%); the mean interval between VL and PKDL was 19 months. A recent longitudinal study in Fulbaria (2015) of 1918 VL patients with active follow-up showed PKDL rates of 10.2% at 36 months (mean 17.6 months; range 4-43 months) after VL treated with 6 x 5 mg/kg Ambisome® (Koert Ritmeijer, MSF, personal communication). Though VL cases are in decline due to extensive programmes conducted by NKEP, PKDL cases are in the rise and VL:PKDL ratio has risen from 1:0.47 to 1:1.21 from 2016 to 2020. In this current situation, elimination of PKDL cases is of crucial importance in the current VL elimination efforts in Bangladesh as well as in the Indian subcontinent.
2. Knowledge gap: Currently there are no satisfactory treatments for any forms of PKDL. Available treatments include pentavalent antimonial sodium stibogluconate (Pentostam, Stibonate) which have been used since the 1940s. Conventional amphotericin B has been used in India for prolonged periods (60 infusions) but this is impractical and requires careful clinical and biochemical monitoring. Both miltefosine and Ambisome® as monotherapy have shown to be effective. However, with the current recommended scheme there are some drawbacks such as the length of the treatment with miltefosine alone (8-12 weeks), toxicity related to it; a high dose Ambisome® (total dose of 20 mg/kg) given frequently in 4 divided dosage often causes adverse events (e.g. pancytopania, hypokalemia, increased creatinine level etc.). There is also the potential risk for development of resistance with miltefosine as monotherapy. Ivermectin has been proven to have a significant leishmanicidal effect by several experimental studies at higher doses without significant toxicity and may offer shorter duration of treatment thus preventing prolonged hospitalization.

   Another possible advantage is reduction of cost. These principles can be applied to PKDL, where the need for an ambulatory treatment with a highly safe, efficacious and user friendly regimen is even more pressing as the patients feel otherwise healthy, except for the rashes.
3. Relevance: This study aims primarily to improve current treatment options. In addition, this will be the first human study ever in PKDL in relation to Ivermectin, in which outcome will be described in clinical, parasitological and immunological terms. Ultimately this study findings will help National Kala-Azar Elimination Program (NKAEP) to adopt specific strategies for elimination of PKDL cases.

Hypothesis (if any): Oral ivermectin in multiple doses is safe and effective for the treatment of PKDL cases.

Objectives: To measure the safety and efficacy of Ivermectin monotherapy regimen (60 mg oral on five consecutive days, for three consecutive months) in treating PKDL patients in Bangladesh.

Methods: This will be a non-control, quasi-experimental, single group, proof of concept, intervention study to assess the safety and efficacy of oral Ivermectin monotherapy (5 x 12 mg daily at a total dose of 60 mg per month for three consecutive months, 180 mg in total) in treating PKDL patients in Bangladesh. In this study we are going to assess whether oral ivermectin in mentioned doses is effective for PKDL treatment or not. All participants will be recruited at SKKRC, Mymensingh with due consent. All patients will be followed up for 6 months since treatment. Cure assessment will be performed. Outcome measures/variables: Safety and efficacy of Ivermectin for PKDL treatment will be determined

ELIGIBILITY:
Inclusion Criteria:

* Confirmed PKDL case of either sex aged more than 5 years,
* Clinically healthy except skin lesions,
* Free from chronic illness
* Normal serum glucose, creatinine and SGPT, Hb ≥ 10 g/dL (male) and 8 g/dL (Female)
* Voluntary participation through informed voluntary written consent.

Exclusion Criteria:

* Incompliance with any inclusion criteria
* Patients who received VL or PKDL treatment within 12 months
* Pregnant / lactating women

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-06-25 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Number of Severe Adverse Events in Participants | Within 3 months following enrollment
  Zero Severe Adverse Events recorded in any of the patients treated with Ivermectin
Number of Participants with Negative PCR Results | Within 12 months after treatment completion
  PCR in Skin samples will be negative for LD-bodies in all the Ivermectin-treated patients

SECONDARY OUTCOMES:
Rate of Reduction in Lesion Number | Within 12 months after treatment completion
  90 % change of PKDL lesions in patients treated with Ivermectin

CONTACTS AND LOCATIONS:
Overall Officials: Shomik Maruf, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b), Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No